CLINICAL TRIAL: NCT01142596
Title: Long-term Extension Trial of Asenapine in Subjects With Schizophrenia (Phase 3 ; Protocol No. P06125)
Brief Title: Long-term Extension Trial of Asenapine in Subjects With Schizophrenia (Study P06125)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Collaborators: Meiji Seika Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P06125; 132324 (Registry Identifier: JAPIC-CTI)
Record Dates: First submitted 2010-06-10; First posted 2010-06-11 (Estimated); Results first posted 2016-05-18 (Estimated); Last update posted 2024-05-28 (Actual); Status verified 2022-02

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — asenapine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Asenapine 5 mg BID (Experimental): Participants continue in the same arm they were on in core trial P06124 (except placebo arm starts 5 mg BID at Week 2) and will be re-randomized after Week 6 to asenapine 5 mg BID or asenapine 10 mg BID, administered open-label for 46 weeks. Open label dose can be adjusted using dose options of 5 and 10 mg BID for efficacy and tolerability
  Interventions: Drug: Asenapine; Drug: Placebo
- Asenapine 10 mg BID (Experimental): Participants continue in the same arm they were on in core trial P06124 (except placebo arm starts 5 mg bid at Week 2) and will be re-randomized after Week 6 to asenapine 5 mg BID or asenapine 10 mg BID, administered open-label for 46 weeks. Open label dose can be adjusted using dose options of 5 and 10 mg BID for efficacy and tolerability
  Interventions: Drug: Asenapine; Drug: Placebo

INTERVENTIONS:
Drug: Asenapine — Asenapine 5 mg sublingual tablet BID, Asenapine 10 mg sublingual tablet BID
  Other Names: SCH 900274
Drug: Placebo — Placebo sublingual tablet BID (first 2 weeks, participants who were in placebo arm of P06124 study only)

SUMMARY:
This is a multi-site, randomized fixed-flexible dose long-term study of asenapine in participants with schizophrenia. The first six weeks of the study will be double-blind and the remainder of the study will be open label. Participants in this study consist of participants who have completed the preceding short-term study (P06124 [NCT01098110]), who meet the inclusion criteria and wish to continue receiving study drug, and whom the investigators have deemed eligible for study participation. Participants who were on placebo twice daily (BID) in core trial P06124 will get placebo for the first 2 weeks then 5 mg asenapine BID for the next 4 weeks of double blind treatment, and will be re-randomized after week 6 to asenapine 5 mg BID or asenapine 10 mg BID. Participants who were on asenapine 5 mg BID in core trial P06124 will be re-randomized after Week 6 to asenapine 5 mg BID or asenapine 10 mg BID. Participants who were on asenapine 10 mg BID in core trial P06124 will be re-randomized after Week 6 to asenapine 5 mg BID or asenapine 10 mg BID. After re-randomization, drug will be administered open-label for 46 weeks. During this period dose is flexible can be adjusted using dose options of 5 and 10 mg BID for efficacy and tolerability.

ELIGIBILITY:
Inclusion Criteria:

* Participant has completed 42-day drug administration in the preceding short-term study (Protocol P06124), has exhibited efficacy (CGI-I at the completion of the preceding short-term study of markedly improved, moderately improved, or slightly improved), has no significant safety problems, and has been judged appropriate for study participation by the investigator.
* Male and female participants. Women who are of childbearing potential (i.e., not surgically sterile or post menopausal for at least 1 year) must use medically acceptable birth control. Medically acceptable birth control includes condoms (male or female) with or without a spermicidal agent, diaphragm or cervical cap with spermicide, medically prescribed IUD, insert or copper-containing IUD, hormone-releasing IUD, systemic hormonal contraceptives, and surgical sterilization (eg, hysterectomy or tubal ligation). Male participants must agree to use condoms during their participation in the study.
* Participant must have been explained the nature of the study by the investigator, and be able to provide written consent prior to the conduct of the tests/observation of the clinical study.

Exclusion Criteria:

* A participant must not have any clinically significant abnormal laboratory, vital sign, physical examination, or electrocardiogram (ECG) findings that, in the investigator's opinion, preclude the participant's participation in the study
* A participant must not have a positive pregnancy test or be planning to become pregnant during the term of the study;
* A participant must not receive antipsychotics, antidepressants, mood stabilizers, anti-epileptics, monoamine oxidase inhibitors, St. John's Wort, antiemetics that are dopamine antagonist, or traditional herbal medication for psychiatric symptoms at the baseline;
* A participant must not be at risk of harming themselves or others, in the investigator's opinion;
* A participant must not have been determined to be unsuitable by an investigator.

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 201 (Actual)
Dates: Start 2010-05-25 (Actual); Primary Completion 2015-04-22 (Actual); Study Completion 2015-04-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kinoshita T, Takekita Y, Hiraoka S, Tamura F, Iwama Y. Long-term safety and efficacy of sublingual asenapine for the treatment of schizophrenia: A phase III extension study with follow-up for 52 weeks (P06125)-Secondary publication. Neuropsychopharmacol Rep. 2023 Sep;43(3):328-337. doi: 10.1002/npr2.12342. Epub 2023 May 25. PMID 37232002

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo/Asenapine: Participants in this group had received double-blind placebo BID in preceding study P06124 (NCT01098110), and continued on same double-blind dose for first 2 weeks of extension study P06125, then took double-blind asenapine 5 mg BID for 4 weeks, after which were re-randomized to open label asenapine 5 or 10 mg BID for 46 weeks. Open label dose could be adjusted using dose options of 5 and 10 mg BID for efficacy and tolerability
- Asenapine 5/10 mg BID: Participants in this group had received double-blind asenapine 5 or 10 mg BID in preceding study P06124, and continued on same double-blind dose for first 6 weeks of extension study P06125, after which were re-randomized to open label asenapine 5 or 10 mg BID for 46 weeks. Open label dose could be adjusted using dose options of 5 and 10 mg BID for efficacy and tolerability
Period: Overall Study
Arm/Group | Placebo/Asenapine | Asenapine 5/10 mg BID
Started | 44 | 157
Completed | 15 | 71
Not Completed | 29 | 86
Not completed — Withdrawal by Subject | 9 | 35
Not completed — Adverse Event | 8 | 35
Not completed — Lack of Efficacy | 5 | 9
Not completed — Lost to Follow-up | 2 | 3
Not completed — Other reason (not specified) | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Placebo/Asenapine: Participants in this group had received double-blind placebo BID in preceding study P06124, and continued on same double-blind dose for first 2 weeks of extension study P06125, then took double-blind asenapine 5 mg BID for 4 weeks, after which were re-randomized to open label asenapine 5 or 10 mg BID for 46 weeks. Open label dose could be adjusted using dose options of 5 and 10 mg BID for efficacy and tolerability
- Total: Total of all reporting groups
Arm/Group | Placebo/Asenapine | Asenapine 5/10 mg BID | Total
Number analyzed (Participants) | 44 | 157 | 201
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.50 (13.39) | 41.82 (11.44) | 41.97 (11.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 79 | 105
  Male | 18 | 78 | 96

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants in Categories of Change in Weight From Study P06124 Baseline to Final Assessment
Description: For each participant, change in weight from preceding 6-week double-blind Study P06124 baseline to the final assessment of extension study P06125 was determined (calculated as final assessment value minus baseline value). Final assessment was last evaluation of participant in study, whether participant completed or did not complete study. Participants were allocated to categories of percentage change from defined baseline to final assessment.
Time Frame: Study P06124 baseline and P06125 study from Day 1 up to Week 52
Population: All participants randomized in study P06125 who received at least one dose of study drug, and had data for measure at study P06124 baseline and study P06125 final assessment
Measure: Number; unit: percentage of participants in category
Arm/Group | Placebo/Asenapine | Asenapine 5/10 mg BID
Number analyzed (Participants) | 31 | 138
percentage of participants in category
  Increase ≥7% | 12.9 | 26.8
  Change within ± 7% | 64.5 | 61.6
  Decrease ≥7% | 22.6 | 11.6

2. Primary Outcome: Percentage of Participants in Categories of Change in Weight From Study P06125 Baseline to Final Assessment
Description: For each participant, change in weight from extension study P06125 baseline to the final assessment of extension study was determined (calculated as final assessment value minus baseline value). Final assessment was last evaluation of participant in study, whether participant completed or did not complete study. Participants were allocated to categories of percentage change from defined baseline to final assessment.
Time Frame: Study P06125 baseline up to Week 52
Population: All participants randomized in study P06125 who received at least one dose of study drug, and had data for measure at study P06125 baseline and final assessment
Measure: Number; unit: percentage of participants in category
Arm/Group | Placebo/Asenapine | Asenapine 5/10 mg BID
Number analyzed (Participants) | 31 | 138
percentage of participants in category
  Increase ≥7% | 22.6 | 23.9
  Change within ± 7% | 64.5 | 62.3
  Decrease ≥7% | 12.9 | 13.8

3. Primary Outcome: Change From Study P06124 Baseline in Body Mass Index (BMI) at Week 52
Description: For each participant, change in BMI from preceding 6-week double-blind Study P06124 baseline to Week 52 of extension study P06125 was determined (calculated as Week 52 value minus baseline value).
Time Frame: Study P06124 baseline and study P06125 Week 52
Population: All participants randomized in study P06125 who received at least one dose of study drug, and had data for measure at study P06124 baseline and study P06125 Week 52
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Placebo/Asenapine | Asenapine 5/10 mg BID
Number analyzed (Participants) | 15 | 70
kg/m^2 | -0.04 (2.83) | 0.91 (2.74)

4. Primary Outcome: Change From Study P06125 Baseline in BMI at Week 52
Description: For each participant, change in BMI from extension study P06125 baseline to Week 52 of extension study was determined (calculated as Week 52 value minus baseline value).
Time Frame: Study P06125 baseline and Week 52
Population: All participants randomized in study P06125 who received at least one dose of study drug, and had data for measure at study P06125 baseline and Week 52
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Placebo/Asenapine | Asenapine 5/10 mg BID
Number analyzed (Participants) | 15 | 70
kg/m^2 | 0.35 (2.48) | 0.75 (2.41)

5. Primary Outcome: Number of Participants With Extrapyramidal Symptoms
Description: This measure reports the overall number of participants with any of a group of adverse events that were defined to represent extrapyramidal symptoms. The number of participants with each of the individual adverse events within this definition is also presented, for terms that occurred in at least one participant. For this measure, all adverse event terms within the Medical Dictionary for Regulatory Activities (MedDRA) Standardized MedDRA Query (SMQ) for "extrapyramidal syndrome" were treated as extrapyramidal symptoms.
Time Frame: Up to 30 days after last dose of study drug (Up to approximately 56 weeks)
Population: All participants randomized in study P06125 who received at least one dose of study drug
Measure: Number; unit: participants
Arm/Group | Placebo/Asenapine | Asenapine 5/10 mg BID
Number analyzed (Participants) | 44 | 157
participants
  Any extrapyramidal symptom | 11 | 34
  Restlessness | 1 | 2
  Akathisia | 2 | 13
  Bradykinesia | 0 | 2
  Dyskinesia | 2 | 3
  Dystonia | 0 | 2
  Extrapyramidal disorder | 2 | 6
  Parkinsonism | 0 | 1
  Tardive dyskinesia | 0 | 1
  Tremor | 4 | 6
  Parkinsonian gait | 1 | 0
  Oromandibular dystonia | 1 | 0
  Blepharospasm | 1 | 0
  Oculogyric crisis | 0 | 1
  Muscle rigidity | 2 | 1
  Muscle tightness | 0 | 1
  Musculoskeletal stiffness | 1 | 2
  Gait disturbance | 0 | 1

6. Primary Outcome: Change From Study P06124 Baseline in Drug-Induced Extrapyramidal Symptoms Scale (DIEPSS) Total Score at Endpoint
Description: Change in DIEPSS Total Score from preceding 6-week double-blind Study P06124 baseline to endpoint assessment of extension study P06125 was determined (calculated as endpoint value minus baseline value). Endpoint assessment was last evaluation of participant for this measure in study, whether participant completed or did not complete study. DIEPSS is a scale, rated by the investigator or rater appointed by the investigator, used to evaluate the severity of drug induced extrapyramidal symptoms occurring during antipsychotic drug treatment. It consists of 9 items: Items 1 through 8 assess individual symptoms; Item 9 is an assessment of global severity. Items 1 through 8 are classified into 4 categories of parkinsonism, akathisia, dystonia and dyskinesia. Each item is rated from 0 (none, normal) to 4 (severe). The Total Score is the sum of scores on Items 1 through 8, with a range from 0 (normal) to 32 (severe). Negative values of change from baseline represent improvement in symptoms.
Time Frame: Study P06124 baseline and P06125 study from Day 1 up to Week 52
Population: All participants randomized in study P06125 who received at least one dose of study drug, and had data for measure at study P06124 baseline and study P06125 endpoint assessment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo/Asenapine | Asenapine 5/10 mg BID
Number analyzed (Participants) | 44 | 153
score on a scale | -0.11 (1.99) | -0.46 (2.54)

7. Primary Outcome: Change From Study P06125 Baseline in DIEPSS Total Score at Endpoint
Description: Change in DIEPSS Total Score from extension study P06125 baseline to the endpoint assessment of extension study was determined (calculated as endpoint value minus baseline value). Endpoint assessment was last evaluation of participant for this measure in study, whether participant completed or did not complete study. DIEPSS is a scale, rated by the investigator or rater appointed by the investigator, used to evaluate the severity of drug induced extrapyramidal symptoms occurring during antipsychotic drug treatment. It consists of 9 items: Items 1 through 8 assess individual symptoms; Item 9 is an assessment of global severity. Items 1 through 8 are classified into 4 categories of parkinsonism, akathisia, dystonia and dyskinesia. Each item is rated from 0 (none, normal) to 4 (severe). The Total Score is the sum of scores on Items 1 through 8, with a range from 0 (normal) to 32 (severe). Negative values of change from baseline represent improvement in symptoms.
Time Frame: Study P06125 baseline up to Week 52
Population: All participants randomized in study P06125 who received at least one dose of study drug, and had data for measure at study P06125 baseline and endpoint assessment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo/Asenapine | Asenapine 5/10 mg BID
Number analyzed (Participants) | 44 | 154
score on a scale | 0.25 (1.57) | -0.03 (1.90)

8. Primary Outcome: Change From Study P06124 Baseline in DIEPSS Item 9 Score at Endpoint
Description: Change in DIEPSS Item 9 (Global) Score from preceding 6-week double-blind Study P06124 baseline to endpoint assessment of extension study P06125 was determined (calculated as endpoint value minus baseline value). Endpoint assessment was last evaluation of participant for this measure in study, whether participant completed or did not complete study. DIEPSS is a scale, rated by the investigator or rater appointed by the investigator, used to evaluate the severity of drug induced extrapyramidal symptoms occurring during antipsychotic drug treatment. It consists of 9 items: Items 1 through 8 assess individual symptoms; Item 9 is an assessment of global severity. Each item is rated from 0 (none, normal) to 4 (severe). Negative values of change from baseline represent improvement in symptoms.
Time Frame: Study P06124 baseline and P06125 study from Day 1 up to Week 52
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo/Asenapine | Asenapine 5/10 mg BID
Number analyzed (Participants) | 44 | 153
score on a scale | 0.14 (0.63) | -0.01 (0.73)

9. Primary Outcome: Change From Study P06125 Baseline in DIEPSS Item 9 Score at Endpoint
Description: Change in DIEPSS Item 9 (Global) Score from extension study P06125 baseline to the endpoint assessment of extension study was determined (calculated as endpoint value minus baseline value). Endpoint assessment was last evaluation of participant for this measure in study, whether participant completed or did not complete study. DIEPSS is a scale, rated by the investigator or rater appointed by the investigator, used to evaluate the severity of drug induced extrapyramidal symptoms occurring during antipsychotic drug treatment. It consists of 9 items: Items 1 through 8 assess individual symptoms; Item 9 is an assessment of global severity. Each item is rated from 0 (none, normal) to 4 (severe). Negative values of change from baseline represent improvement in symptoms.
Time Frame: Study P06125 baseline up to Week 52
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo/Asenapine | Asenapine 5/10 mg BID
Number analyzed (Participants) | 44 | 154
score on a scale | 0.18 (0.69) | -0.02 (0.62)

10. Primary Outcome: Change From Study P06124 Baseline in Glycosylated Hemoglobin (HbA1c) at Week 52
Description: For each participant, change in HbA1c from preceding 6-week double-blind Study P06124 baseline to Week 52 of extension study P06125 was determined (calculated as Week 52 value minus baseline value).
Time Frame: Study P06124 baseline and study P06125 Week 52
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percentage of HbA1c
Arm/Group | Placebo/Asenapine | Asenapine 5/10 mg BID
Number analyzed (Participants) | 15 | 68
percentage of HbA1c | -0.09 (0.44) | -0.02 (0.82)

11. Primary Outcome: Change From Study P06125 Baseline in HbA1c at Week 52
Description: For each participant, change in HbA1c from extension study P06125 baseline to Week 52 of extension study was determined (calculated as Week 52 value minus baseline value).
Time Frame: Study P06125 baseline and Week 52
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percentage of HbA1c
Arm/Group | Placebo/Asenapine | Asenapine 5/10 mg BID
Number analyzed (Participants) | 15 | 69
percentage of HbA1c | 0.21 (0.36) | 0.12 (1.02)

12. Primary Outcome: Change From Study P06124 Baseline in Fasting Glucose at Week 52
Description: For each participant, change in fasting glucose from preceding 6-week double-blind Study P06124 baseline to Week 52 of extension study P06125 was determined (calculated as Week 52 value minus baseline value).
Time Frame: Study P06124 baseline and study P06125 Week 52
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo/Asenapine | Asenapine 5/10 mg BID
Number analyzed (Participants) | 14 | 64
mmol/L | 0.37 (1.00) | 0.28 (1.93)

13. Primary Outcome: Change From Study P06125 Baseline in Fasting Glucose at Week 52
Description: For each participant, change in fasting glucose from extension study P06125 baseline to Week 52 of extension study was determined (calculated as Week 52 value minus baseline value).
Time Frame: Study P06125 baseline and Week 52
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo/Asenapine | Asenapine 5/10 mg BID
Number analyzed (Participants) | 14 | 65
mmol/L | 0.60 (1.79) | 0.00 (2.16)

14. Primary Outcome: Change From Study P06124 Baseline in Insulin at Week 52
Description: For each participant, change in insulin from preceding 6-week double-blind Study P06124 baseline to Week 52 of extension study P06125 was determined (calculated as Week 52 value minus baseline value).
Time Frame: Study P06124 baseline and study P06125 Week 52
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: μIU/mL
Arm/Group | Placebo/Asenapine | Asenapine 5/10 mg BID
Number analyzed (Participants) | 14 | 69
μIU/mL | 4.06 (16.27) | 2.24 (16.06)

15. Primary Outcome: Change From Study P06125 Baseline in Insulin at Week 52
Description: For each participant, change in insulin from extension study P06125 baseline to Week 52 of extension study was determined (calculated as Week 52 value minus baseline value).
Time Frame: Study P06125 baseline and Week 52
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: μIU/mL
Arm/Group | Placebo/Asenapine | Asenapine 5/10 mg BID
Number analyzed (Participants) | 14 | 69
μIU/mL | -5.61 (28.89) | 0.56 (17.88)

16. Primary Outcome: Change From Study P06124 Baseline in Prolactin at Week 52
Description: For each participant, change in prolactin from preceding 6-week double-blind Study P06124 baseline to Week 52 of extension study P06125 was determined (calculated as Week 52 value minus baseline value).
Time Frame: Study P06124 baseline and study P06125 Week 52
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: μg/L
Arm/Group | Placebo/Asenapine | Asenapine 5/10 mg BID
Number analyzed (Participants) | 15 | 70
μg/L | -37.46 (68.83) | -20.98 (47.14)

17. Primary Outcome: Change From Study P06125 Baseline in Prolactin at Week 52
Description: For each participant, change in prolactin from extension study P06125 baseline to Week 52 of extension study was determined (calculated as Week 52 value minus baseline value).
Time Frame: Study P06125 baseline and Week 52
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: μg/L
Arm/Group | Placebo/Asenapine | Asenapine 5/10 mg BID
Number analyzed (Participants) | 15 | 70
μg/L | 10.91 (20.58) | -1.59 (17.22)

18. Primary Outcome: Number of Participants With Serious Adverse Events (AEs)
Description: An AE is defined as any untoward medical occurrence in a participant administered study drug and which does not necessarily have to have a causal relationship with the study drug. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with study drug administration, whether or not considered related to study drug. A serious AE (SAE) is any AE occurring at any dose that results in death, is life-threatening, results in hospitalization or prolongation of hospitalization, results in persistent or significant disability/incapacity, or is a congenital anomaly/birth defect. In addition, an important medical event that may not result in death, be life-threatening, or require hospitalization may be considered an SAE when it may jeopardize the participant and may require medical or surgical intervention to prevent one of the outcomes listed in this definition.
Time Frame: Up to 30 days after last dose of study drug (Up to approximately 56 weeks)
Population: All participants randomized in study P06125 who received at least one dose of study drug
Measure: Number; unit: participants
Arm/Group | Placebo/Asenapine | Asenapine 5/10 mg BID
Number analyzed (Participants) | 44 | 157
participants | 5 | 32

19. Primary Outcome: Number of Participants With Non-serious AEs
Description: An AE is defined as any untoward medical occurrence in a participant administered study drug and which does not necessarily have to have a causal relationship with the study drug. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with study drug administration, whether or not considered related to study drug. This measure presents the number of participants with at least one AEs that was non-serious (i.e., was not determined to be an SAE).
Time Frame: Up to 30 days after last dose of study drug (Up to approximately 56 weeks)
Population: All participants randomized in study P06125 who received at least one dose of study drug
Measure: Number; unit: participants
Arm/Group | Placebo/Asenapine | Asenapine 5/10 mg BID
Number analyzed (Participants) | 44 | 157
participants | 40 | 131

20. Primary Outcome: Percentage of Participants With Abnormalities on Electrocardiogram (ECG) at Study P06124 Baseline, Study P06125 Baseline and Week 52
Description: The percentage of participants with abnormal ECG findings is reported for three time points: 6-week double-blind study P06124 baseline, extension study P06125 baseline and extension study Week 52.
Time Frame: Study P06124 baseline and P06125 study baseline and Week 52
Population: All participants randomized in study P06125 who received at least one dose of study drug
Measure: Number; unit: percentage of participants
Arm/Group | Placebo/Asenapine | Asenapine 5/10 mg BID
Number analyzed (Participants) | 44 | 157
percentage of participants
  P06124 baseline (N = 43, 153) | 41.9 | 24.8
  P06125 baseline (N = 44, 156) | 34.1 | 26.9
  Week 52 (N = 14, 70) | 42.9 | 25.7

21. Primary Outcome: Number of Participants Who Took Antiparkinsonian Drugs
Description: This measure presents the number of participants who used antiparkinsonian drugs started on or after the start of study treatment in extension study P06125. Antiparkinsonian drugs were defined as those categorized into the N04 code (antiparkinson drugs) of the World Health Organization (WHO) Anatomical Therapeutic Chemical (ATC) classification system.
Time Frame: P06125 study from Day 1 up to Week 52
Population: All participants randomized in study P06125 who received at least one dose of study drug
Measure: Number; unit: participants
Arm/Group | Placebo/Asenapine | Asenapine 5/10 mg BID
Number analyzed (Participants) | 44 | 157
participants
  Any antiparkinsonian drug | 12 | 40
  Biperiden | 4 | 8
  Biperiden hydrochloride | 3 | 16
  Procyclidine | 2 | 1
  Trihexyphenidyl | 0 | 3
  Trihexyphenidyl hydrochloride | 1 | 7
  Benzatropine mesilate | 4 | 5

22. Primary Outcome: Median Time to Loss of Effect in Responders
Description: Median time to loss of effect from P06125 extension study baseline was estimated using Kaplan-Meier product-limit method. Result reported in Responders, participants with ≥30% decrease from study P06124 baseline in Positive and Negative Syndrome Scale (PANSS, schizophrenia symptom scale) Total Score at the end of study P06124. Investigator or subinvestigator was to determine whether the study drug failed to maintain effect based on occurrence of any of the following: 1) Increase in PANSS Total Score ≥30% from P06125 extension study baseline, 2) Determination that participant's schizophrenic symptomatology had deteriorated requiring one or more of defined interventions (add new antipsychotic drug, increase in level of psychiatric outpatient care, or hospitalization/increase in level of hospitalization for psychiatric need), 3) Clinical Global Impression-Severity (CGI-S) score ≥6, 4) Discontinuation from study because of lack of efficacy, 5) AE/SAE of worsening of schizophrenia.
Time Frame: P06124 study baseline and Day 42, and P06125 study from Day 1 up to Week 52
Population: All participants randomized in study P06125 who received at least one dose of study drug, had PANSS measurement at P06125 baseline and at least one post-baseline PANSS measurement, and were study P06124 Responders
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Placebo/Asenapine | Asenapine 5/10 mg BID
Number analyzed (Participants) | 25 | 101
days | 357.0 [18.0 to NA] — Data were insufficient to calculate upper 95% confidence interval limit | 177.0 [91.0 to NA] — Data were insufficient to calculate upper 95% confidence interval limit

23. Primary Outcome: Median Time to Loss of Effect in Non-Responders
Description: Median time to loss of effect from P06125 extension study baseline was estimated using Kaplan-Meier product-limit method. Result reported in Non-Responders, participants without ≥30% decrease from study P06124 baseline in PANSS Total Score at the end of study P06124. Investigator or subinvestigator was to determine whether the study drug failed to maintain effect based on occurrence of any of the following: 1) Increase in PANSS Total Score ≥30% from P06125 extension study baseline, 2) Determination that participant's schizophrenic symptomatology had deteriorated requiring one or more of defined interventions (add new antipsychotic drug, increase in level of psychiatric outpatient care, or hospitalization/increase in level of hospitalization for psychiatric need), 3) Clinical Global Impression-Severity (CGI-S) score ≥6, 4) Discontinuation from study because of lack of efficacy, 5) AE/SAE of worsening of schizophrenia.
Time Frame: P06124 study baseline and Day 42, and P06125 study from Day 1 up to Week 52
Population: All participants randomized in study P06125 who received at least one dose of study drug, had PANSS measurement at P06125 baseline and at least one post-baseline PANSS measurement, and were study P06124 Non-Responders
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Placebo/Asenapine | Asenapine 5/10 mg BID
Number analyzed (Participants) | 19 | 52
days | 53.0 [14.0 to NA] — Data were insufficient to calculate upper 95% confidence interval limit | 368.0 [229.0 to NA] — Data were insufficient to calculate upper 95% confidence interval limit

ADVERSE EVENTS:
Time Frame: Up to 30 days after last dose of study drug (Up to approximately 56 weeks)
Arm/Group | Placebo/Asenapine | Asenapine 5/10 mg BID
Serious Adverse Events (participants affected / at risk) | 5/44 | 32/157
Other Adverse Events (participants affected / at risk) | 34/44 | 98/157
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo/Asenapine (N=44) | Asenapine 5/10 mg BID (N=157)
Gastritis (Gastrointestinal disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Polydipsia (Metabolism and nutrition disorders) | 0 | 1
Water intoxication (Metabolism and nutrition disorders) | 0 | 1
Muscle rigidity (Musculoskeletal and connective tissue disorders) | 0 | 1
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neuroleptic malignant syndrome (Nervous system disorders) | 0 | 1
Somnolence (Nervous system disorders) | 0 | 1
Abnormal behaviour (Psychiatric disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1
Completed suicide (Psychiatric disorders) | 1 | 0
Depressed mood (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 0 | 1
Irritability (Psychiatric disorders) | 0 | 1
Panic attack (Psychiatric disorders) | 0 | 1
Restlessness (Psychiatric disorders) | 0 | 1
Schizophrenia (Psychiatric disorders) | 4 | 22
Sleep disorder (Psychiatric disorders) | 1 | 0
Stress (Psychiatric disorders) | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 3
Hypotension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo/Asenapine (N=44) | Asenapine 5/10 mg BID (N=157)
Palpitations (Cardiac disorders) | 3 | 2
Constipation (Gastrointestinal disorders) | 4 | 12
Hypoaesthesia oral (Gastrointestinal disorders) | 4 | 1
Stomatitis (Gastrointestinal disorders) | 4 | 2
Nasopharyngitis (Infections and infestations) | 6 | 34
Aalanine aminotranferase increased (Investigations) | 3 | 8
Weight increased (Investigations) | 7 | 17
Hyperlipidaemia (Metabolism and nutrition disorders) | 3 | 3
Akathisia (Nervous system disorders) | 2 | 13
Dizziness (Nervous system disorders) | 2 | 9
Headache (Nervous system disorders) | 9 | 9
Somnolence (Nervous system disorders) | 5 | 17
Tremor (Nervous system disorders) | 4 | 6
Insomnia (Psychiatric disorders) | 2 | 12
Schizophrenia (Psychiatric disorders) | 6 | 17
Dysmenorrhea (Reproductive system and breast disorders) | 3 | 1
Eczema (Skin and subcutaneous tissue disorders) | 3 | 5
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
It is planned to first publish/present trial results together with the other sites, unless permission is obtained from Sponsor to publish separate results. Sponsor must be able to review all proposed results communications regarding study 45 days prior to submission for publication/presentation. If there is disagreement concerning appropriateness of the materials, Investigator and Sponsor must meet to make a good faith effort to discuss/resolve disagreement prior to submission for publication.